CLINICAL TRIAL: NCT00246974
Title: An Open Randomised Phase II Study Of Gemcitabine Plus Cisplatin +/- Concomitant or Sequential ZD1839 in Patients With Advanced or Metastatic Transitional Cell Carcinoma of the Urothelium
Brief Title: Phase II Gemcitabine + Cisplatin +/- Iressa Bladder CCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1839IL/0063; D7913L00063
Record Dates: First submitted 2005-10-31; First posted 2005-11-01 (Estimated); Last update posted 2008-10-15 (Estimated); Status verified 2008-10

CONDITIONS: Bladder Cancer
Keywords: bladder cancer; Transitionel cell cancer of the urothelium
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Gemcitabine; Cisplatin; Gefitinib

ARMS (2):
- 1 (Active Comparator): Cisplatin + Gemcitabin
  Interventions: Drug: Gemcitabine; Drug: Cisplatin
- 2 (Experimental): Cisplatin + Gemcitabin + Gefitinib
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Drug: Gefitinib

INTERVENTIONS:
Drug: Gemcitabine — intravenous
Drug: Cisplatin — intravenous
Drug: Gefitinib — oral
  Other Names: Iressa; ZD1839
  Arms: 2

SUMMARY:
The primary objective of the study is to assess the activity of ZD1839 250 mg once daily in addition to the standard chemotherapy in patients with advanced or metastatic transitional cell carcinoma of the urothelium by estimating the time to progression.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically-confirmed transitional cell carcinoma of the urothelium
* Locally advanced or metastatic disease
* At least one measurable lesion as defined by RECIST
* Chemotherapy-naiv

Exclusion Criteria:

* Previous chemotherapy or other systemic antitumour therapy
* Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of basal cell carcinoma, cervical cancer in situ or locally limited prostate cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2003-05; Primary Completion 2007-10 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Time to progression (TTP)

SECONDARY OUTCOMES:
1. Response rate
2. Overall survival time
3. Time to treatment failure
4. Disease control rate
5. Duration of response
6. Safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Iressa Medical Science Director, MD, Study Director — AstraZeneca
Locations (14):
- Germany (14):
  - Research Site, Aachen
  - Research Site, Augsburg
  - Research Site, Berlin
  - Research Site, Dresden
  - Research Site, Freiburg im Breisgau
  - Research Site, Halle
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Kassel
  - Research Site, Mainz
  - Research Site, Mannheim
  - Research Site, Münster
  - Research Site, Tübingen
  - Research Site, Ulm